CLINICAL TRIAL: NCT01770691
Title: Preliminary Performance Study of the New TIPI Device in the Prevention of Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIPI 004
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TIPI vaginal pessary (Experimental): Each subject will use different SMD'S (Slightly modified designs) of the TIPI vaginal pessary. Not all subjects will use all types of SMD's
  Interventions: Device: TIPI vaginal pessary

INTERVENTIONS:
Device: TIPI vaginal pessary — TIPI vaginal pessary G3 model, and TIPI SMD's

SUMMARY:
Stress urinary incontinence (SUI) is most prevalent among women. SUI is characterized by loss of urine from increased abdominal pressures caused by coughing, laughing, sneezing, running, lifting or walking. SUI cause women to avoid routine physical activities, thus detracting significantly from their quality of life.

The purpose of this study is to evaluate the performance of new designs of the TIPI device, a conservative, disposable, treatment for temporary management of SUI.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 to 60 years
* Had ≥ 1 deliveries
* Suffering from genuine stress urinary incontinence confirmed by urodynamic testing (Urodynamic stress urinary incontinence) and normal voiding without abnormal residual urine
* Baseline PWG (no usage of TIPI device) ≥ 6gr/8hrs
* Average reduction of urinary incontinence of at least 70% following 3 days usage of the cleared TIPI G3 device
* The patient has the ability to understand the nature of the study and give her consent by signing a written informed consent form.
* Successful experience with the use of vaginal tampons
* Willing to undergo urodynamic investigation
* Normal pap smear within past 24 months
* Patient is able and agrees to arrive to the study site area for a period of about 4-6 hours during 6-12 non consequent study days.

Exclusion Criteria:

* Patient is pregnant, or suspected to be pregnant or is planning to be pregnant during the course of the study
* Patients with present or suspected urinary infection
* Patients with present or suspected vaginal infection
* Severely atrophic vagina
* Women who did not manage to insert a vaginal tampon, for any reason, in the past
* Abnormal vaginal bleeding
* Patient is currently participating in another clinical study that may directly or indirectly affect the results of this study
* Was/is being treated for urinary incontinence by other means such as medications, surgical intervention etc. that might influence study results
* Vaginal wall prolapse of any type reaching the level of the introitus (grade 2)
* Co-morbid condition(s) that could limit the patient's ability to participate in the study, or impact the scientific integrity of the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elan Ziv, MD, OBGYN, Principal Investigator — Urodynamic Unit, Assuta Medical Centers, Tel Aviv, Israel
Locations (1):
- Urodynamic Unit, Assuta Medical Centers, Tel Aviv, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- TIPI Vaginal Pessary: Each subject will use different SMD'S (Slightly modified designs) of the TIPI vaginal pessary. Not all subjects will use all SMD'S
  TIPI vaginal pessary: TIPI vaginal pessary G3 model, and TIPI SMD's
Period: Overall Study
Arm/Group | TIPI Vaginal Pessary
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- TIPI Vaginal Pessary: Each subject will use different SMD'S (Slightly modified designs) of the TIPI vaginal pessary.
  TIPI vaginal pessary: TIPI vaginal pessary G3 model, and TIPI SMD's
Arm/Group | TIPI Vaginal Pessary
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: Years] | 54.67 [47.1 to 62.9]
Sex/Gender, Customized [Number; unit: Participants]
  Female | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Pad Weight Gain (PWG) Change
Description: All eligible subjects underwent a 3-day Pad period to establish baseline Average PWG. During this period, pre-weighed pads were worn for 8 hours a day and subjects were asked to perform predefined physical activities and drink a certain amount of liquid, daily. Pads were collected and weighed in the clinic to determine baseline urine leakage. Subjects then used SMDs or the cleared TIPI (G3) with pads for up to 8 hours. The average PWG tests results with the TIPI devices were compared to the average PWG 8 hrs test without the device and were presented as percentages.
  The efficacy endpoint for the study was mean percent change of PWG using a certain device compared to the values obtained at the baseline period, as calculated by the following formula:
  % Reduction = 1-(Device/Baseline )*100
  Where, Device = the average pad weight gain (PWG) during device usage. Baseline = the average pad weight gain (PWG) during the days of baseline period.
Time Frame: up to 8 hours of use
Measure: Mean (Standard Deviation); unit: Mean percentage of PWG change
Groups:
- SMD 12 2008: 5 subjects used SMD 12 for up to 8 hours during 2008
- SMD 12 2009: 6 subjects used SMD 12 for up to 8 hours during 2009
- SMD 9: 7 subjects used SMD 9 for up to 8 hours
- Cleared TIPI Device (G3): 7 subjects used the cleared TIPI G3 for up to 8 hours
Arm/Group | SMD 12 2008 | SMD 12 2009 | SMD 9 | Cleared TIPI Device (G3)
Number analyzed (Participants) | 5 | 6 | 7 | 7
Mean percentage of PWG change | 90.8 (16.9) | 98.5 (1.35) | 99.3 (0.61) | 89.3 (17.9)

ADVERSE EVENTS:
Arm/Group | TIPI Vaginal Pessary
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIPI Vaginal Pessary (N=7)
Spotting (General disorders) | 3 (6) — Six (6) spotting (small blood spots detected on the TIPI cover after removal) events out of 55 usages were recored with the main TIPI SMDs. All adverse events were considered to be mild, minimal and temporary, and resolved with no sequelae.
Spotting (General disorders) | 2 (5) — Five (5) spotting (small blood spots detected on the TIPI cover after removal) events out of 42 usages were recorded with the cleared TIPI device. All adverse events were considered to be mild, minimal and temporary, and resolved with no sequela.
Discomfort (General disorders) | 2 (2) — Two (2) discomfort events out of 42 usages of the cleared TIPI device were recorded. All adverse events were considered to be mild, minimal and temporary, and resolved with no sequela.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes